CLINICAL TRIAL: NCT03217838
Title: A Phase I/II, Open-Label, Multicentre 2-Part Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of AZD2811 as Monotherapy or in Combination in Treatment-Naïve or Relapsed/Refractory Acute Myeloid Leukaemia Patients Not Eligible for Intensive Induction Therapy.
Brief Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of AZD2811 Nanoparticles as Monotherapy or in Combination in Acute Myeloid Leukemia Participants.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: strategic decision
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6130C00003; HEMREF 41 (Other: Sarah Cannon Development Innovations, LLC)
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukaemia
Keywords: AML; Acute Myeloid Leukaemia; AZD2811; AZD1152; AZD1152 hQPA; barasertib; azacitidine; VIDAZA®; venetoclax; VENCLEXTA®
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — AZD2811; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Group 1 Arm A (AZD2811 Dose 1) (Experimental): Participants with AML will receive intevenous (IV) infusion of AZD2811 Dose 1 on Days 1 and 4 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm A (AZD2811 Dose 2) (Experimental): Participants with AML and myelodysplastic syndrome (MDS) will receive IV infusion of AZD2811 Dose 2 on Days 1 and 4 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm A (AZD2811 Dose 3) (Experimental): Participants with AML and MDS will receive IV infusion of AZD2811 Dose 3 on Days 1 and 4 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm A (AZD2811 Dose 4) (Experimental): Participants with AML and MDS will receive IV infusion of AZD2811 Dose 4 on Days 1 and 4 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm A (AZD2811 Dose 5) (Experimental): Participants with AML will receive IV infusion of AZD2811 Dose 5 on Days 1 and 4 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm B (AZD2811 Dose 2) (Experimental): Participants with AML will receive IV infusion of AZD2811 Dose 2 on Days 1, 4, 15, and 18 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 1 Arm B (AZD2811 Dose 6) (Experimental): Participants with AML will receive IV infusion of AZD2811 Dose 6 on Days 1, 4, 15, and 18 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811
- Group 2 Arm A (AZD2811 Dose 3 + Azacitidine 75 mg/m^2) (Experimental): Participants with AML and MDS will receive Azacitidine 75 mg/m^2 of body surface area (BSA) by subcutaneous (SC) injection or IV infusion prior to the start of AZD2811 infusion on Days 1 through 7 or for 5 consecutive weekdays (Days 1 through 5) with treatment holidays on the 2 weekend days (Days 6 and 7), and the remaining azacitidine dosing will be administered on the first 2 weekdays of the 2nd week (Days 8 and 9) of each 28-day cycle. Participants will receive IV infusion of AZD2811 Dose 3 on Days 1 and 4 of each 28-day cycle. Participants will receive the study treatment until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Azacitidine
- Group 2 Arm A (AZD2811 Dose 4 + Azacitidine 75 mg/m^2) (Experimental): Participants with AML will receive Azacitidine 75 mg/m^2 of BSA by SC injection or IV infusion prior to the start of AZD2811 infusion on Days 1 through 7 or for 5 consecutive weekdays (Days 1 through 5) with treatment holidays on the 2 weekend days (Days 6 and 7), and the remaining azacitidine dosing will be administered on the first 2 weekdays of the 2nd week (Days 8 and 9) of each 28-day cycle. Participants will receive IV infusion of AZD2811 Dose 4 on Days 1 and 4 of each 28-day cycle. Participants will receive the treatment until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Azacitidine
- Group 2 Arm B (AZD2811 Dose 2 + Azacitidine 75 mg/m^2) (Experimental): Participants with AML will receive Azacitidine 75 mg/m^2 of BSA by SC injection or IV infusion prior to the start of AZD2811 infusion on Days 1 through 7 or for 5 consecutive weekdays (Days 1 through 5) with treatment holidays on the 2 weekend days (Days 6 and 7), and the remaining azacitidine dosing will be administered on the first 2 weekdays of the 2nd week (Days 8 and 9) of each 28-day cycle. Participants will receive IV infusion of AZD2811 Dose 2 on Days 1, 4, 15, and 18 of each 28-day cycle. Participants will receive the treatment until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Azacitidine
- Group 2 Arm B (AZD2811 Dose 6 + Azacitidine 75 mg/m^2) (Experimental): Participants with AML will receive Azacitidine 75 mg/m^2 of BSA by SC injection or IV infusion prior to the start of AZD2811 infusion on Days 1 through 7 or for 5 consecutive weekdays (Days 1 through 5) with treatment holidays on the 2 weekend days (Days 6 and 7), and the remaining azacitidine dosing will be administered on the first 2 weekdays of the 2nd week (Days 8 and 9) of each 28-day cycle. Participants will receive IV infusion of AZD2811 Dose 6 on Days 1, 4, 15, and 18 of each 28-day cycle. Participants will receive the treatment until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Azacitidine
- Group 3 Arm A (AZD2811 Dose 2 + Venetoclax 200 mg) (Experimental): Participants with AML will receive IV infusion of AZD2811 Dose 2 on Days 1 and 4 of each 28-day cycle and venetoclax 100 mg orally (PO) on Day 1 and 200 mg PO from Days 2 to 28 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Venetoclax
- Group 3 Arm A (AZD2811 Dose 2 + Venetoclax 400 mg) (Experimental): Participants with AML will receive IV infusion of AZD2811 Dose 2 on Days 1 and 4 of each 28-day cycle and venetoclax 100 mg orally (PO) on Day 1, 200 mg PO on Day 2, and 400 mg PO from Days 3 to 28 of each 28-day cycle until disease progression, unacceptable toxicity, or the decision to discontinue treatment by the participant or the study physician, whichever occurs first.
  Interventions: Drug: AZD2811; Drug: Venetoclax

INTERVENTIONS:
Drug: AZD2811 — AZD2811 will be administered by IV infusion with the specified dose level as reported in arms in 28-day cycles.
  Other Names: AZD1152 hQPA; AZD1152 hydroxyl-quinazoline pyrazole anilide
Drug: Azacitidine — Azacitidine is supplied in vials of 25 mg/mL powder for suspension for injection. After reconstitution, each vial contains a maximum of 100 mg. Participants should be pre-medicated for nausea and vomiting according to institutional standards before receiving azacitidine. Participants will receive 75 mg/m² on Days 1 through 7 or for 5 consecutive weekdays with rest on the 2 weekend days, and azacitidine dosing the first 2 weekdays of the next week of each 28-day cycle.
  Other Names: Vidaza (TM)
  Arms: Group 2 Arm A (AZD2811 Dose 3 + Azacitidine 75 mg/m^2); Group 2 Arm A (AZD2811 Dose 4 + Azacitidine 75 mg/m^2); Group 2 Arm B (AZD2811 Dose 2 + Azacitidine 75 mg/m^2); Group 2 Arm B (AZD2811 Dose 6 + Azacitidine 75 mg/m^2)
Drug: Venetoclax — Venetoclax (VENCLEXTA®) is approved by the FDA for use in combination with azacitidine, or decitabine, or low-dose cytarabine for the treatment of newly-diagnosed AML in adults who are age 75 years or older, or who have comorbidities that preclude use of intensive induction chemotherapy. Venetoclax is planned to be given at a dose of 100 mg orally (PO) on Day 1 and 200 mg (PO) on Days 2- 28 of each 28-day cycle or 100 mg orally (PO) on Day 1, 200 mg PO on Day 2, and 400 mg PO from Days 3 to 28 of each 28-day cycle. The third participant in Group 3 Arm A will only be enrolled after the first 2 participants will receive ≥2 weeks of treatment and have shown no evidence of toxicity observed to be compatible with a DLT.
  Other Names: Venclexta (TM)
  Arms: Group 3 Arm A (AZD2811 Dose 2 + Venetoclax 200 mg); Group 3 Arm A (AZD2811 Dose 2 + Venetoclax 400 mg)

SUMMARY:
This is a Phase I/II clinical study to determine the maximum tolerated dose (MTD), and schedule, safety, tolerability, pharmacokinetics, and pharmacodynamics of AZD2811 monotherapy or with combination agent(s) in relapsed/refractory acute myeloid leukaemia (AML) participants or treatment-naïve AML participants not eligible for intensive induction therapy. In addition, the study will explore the potential clinical activity by assessing anti-tumour activity in participants. The study was terminated early as a result of AstraZeneca's strategic review across the AZD2811 programme. Part A data were collected for initial cohorts; the MTD/recommended Phase 2 dose (RP2D) dose and schedule of AZD2811 monotherapy or with combination agents were not determined. Part B of the study was not initiated

DETAILED DESCRIPTION:
This is a Phase I/II clinical study to determine the MTD and schedule, safety, tolerability, pharmacokinetics, and pharmacodynamics of AZD2811 monotherapy or with combination agent(s) in relapsed/refractory AML participants or treatment-naïve AML participants not eligible for intensive induction therapy. The study will also explore the potential clinical activity by assessing anti-tumour activity in participants. The study will be conducted in two parts, designated Part A, dose escalation, and Part B, dose expansion. Participants will be enrolled in either Part A or Part B according to the Investigator's judgment of the most appropriate treatment for the individual participant and slot availability.

Part A - Dose Escalation

Approximately 48 evaluable treatment-naïve AML participants not eligible for intensive induction therapy or relapsed/refractory AML participants will be enrolled in Arm 1 and Arm 2 of the monotherapy escalation in Part A of this study.

The dose escalation and de-escalation plan for evaluating AZD2811 will follow the Bayesian Adaptive Design scheme which combines prior expectations about the dose toxicity relationship and applies the data at the end of each cohort to recommend a dose and schedule for the next cohort. The total number of participants will depend upon the number of dose escalations, de-escalations, and schedule changes necessary. At least 3 and up to 6 evaluable participants will be required for each dose cohort.

Part A Group 1, Arm A - Day 1 and 4 Monotherapy Dose Escalation:

Participants will receive a single 2- or 4- hour IV infusion on Day 1 and Day 4 of each 28-day cycle. Dosing frequency and schedule may be adjusted during the study on the basis of emerging safety and pharmacokinetic data. Approximately 22 participants will be enrolled.

Part A Group 1, Arm B - Day 1, 4, 15, and 18 Monotherapy Dose Escalation:

A Day 1, 4, 15, and 18 every 4 weeks or 28 days (Q4W) schedule will be investigated in addition to the Day 1 and 4 Q4W schedule. The proposed starting dose for this schedule is 300 mg/infusion AZD2811 on Day 1, 4, 15 and 18 (i.e. cumulative dose 1200 mg/Q4W). This starting dose is less than daily doses shown to be tolerated in the AML setting, and the cumulative cycle dose/Q4W does not exceed the highest dose shown to be tolerated (600 mg/infusion Day 1, 4 cumulative 1200 mg Q4W). Approximately 18 participants will be enrolled.

Combination Escalation:

AZD2811 can be escalated (in the combination setting) independent of the monotherapy dose explored, after thorough examination of the available safety data. The combination therapy exploration will not impact the dose to be further explored in the monotherapy setting nor will the monotherapy impact the dose in the combination setting. As such, the number of cohorts in the monotherapy setting can differ from the number of cohorts in the combination setting. The safety observations of the monotherapy will be considered by the Safety Review Committee (SRC) in the overall decision-making process for subsequent dose exploration decision.

A rolling 6 design will be applied to both of the AZD2811 and combination arms. The rolling 6 method allows accrual of 3 to 6 participants concurrently onto a dose level based on the numbers of participants who are currently enrolled and evaluable, who experience a dose-limiting toxicity (DLT), and who remain at risk of developing a DLT.

Part A Group 2 Arm A - Day 1 and 4 Azacitidine Combination Escalation:

A starting dose of 400 mg of AZD2811 will be used for investigation in combination with the standard dose of the hypomethylating agent (HMA) azacitidine. In this dose escalation part, approximately 12-15 evaluable treatment-naïve AML participants not eligible for intensive induction therapy or relapsed/refractory AML will be enrolled and dosed in ascending doses of AZD2811 and standard dose of azacitidine at 75 mg/m² of body surface area subcutaneously (SC) in all territories or optionally/alternatively by IV in the United States (US) as per national prescribing information.

Part A Group 2 Arm B - Day 1, 4, 15, and 18 Azacitidine Combination Dose Escalation

In order to increase dose intensity during the 4 week cycle, and improve efficacy in the combination setting, AZD2811 will also be explored on the Days 1, 4, 15 and 18 schedule in the azacitidine combination and start at a lower daily dosage that has been shown to be safe while administered every 28 days. The proposed starting dose for this schedule is 300 mg/infusion AZD2811 on Day 1, 4, 15 and 18 (i.e., cumulative dose per 28 days is 1200 mg/Q4W) and standard dose and use of azacitidine 75 mg/m² of body surface area SC in all territories or optionally/alternatively by IV in the US as per national prescribing information. Approximately 18 participants will be enrolled.

Venetoclax Combination:

Approximately 18-21 evaluable relapsed/refractory AML participants will be enrolled and dosed with AZD2811 and venetoclax. In cohort 1v, AZD2811 will be administered at 200 mg IV on Days 1 and 4 every 28 days (Q4W) and venetoclax will be given 100 mg orally (PO) on Day 1 and 200 mg (PO) with a meal and water on Days 2- 28 for the 1st cycle. The third participant in cohort 1 (AZD2811 at 200 mg) will only be enrolled after the first 2 participants have received ≥ 2 weeks of treatment and have shown no evidence of toxicity observed to be compatible with a DLT, and further dose escalations of AZD2811 will occur at the discretion of the SRC.

The dose of AZD2811 can be escalated (in the combination setting) independent of the monotherapy dose explored, after thorough examination of the available safety data of the current and the previous cohorts. The combination therapy exploration will not impact the dose further explored in the monotherapy setting nor will the monotherapy impact the dose in the combination setting. As such, the number of cohorts in the monotherapy setting can differ from the number of cohorts in the combination setting. The safety observations of the monotherapy will be considered by the SRC in the overall decision-making process for subsequent dose exploration decision.

Part A Group 3 Arm A - Day 1 and 4 Venetoclax Combination Dose Escalation

In Group 3 Arm A, AZD2811 is planned to be administered at 200 mg IV on Day 1 and Day 4 every 28 days (Q4W) and venetoclax is planned to be given (with a meal and water) at a dose of 100 mg orally (PO) on Day 1 and ramping up to 200 mg (PO) on Days 2-28 for the 1st cycle. The third participant in cohort 1 (AZD2811 at 200 mg) will only be enrolled after the first 2 participants have received ≥2 weeks of treatment and have shown no evidence of toxicity observed to be compatible with a DLT.

Further dose escalations of AZD2811 in Group 3 Arm A will occur at the discretion of the SRC.

Part A Group 3 Arm B - Day 1, 4, 15, and 18 Venetoclax Combination Dose Escalation

If data from Groups 1 and/or 2 suggest that participants could benefit from a more intense AZD2811 dosing regimen, a schedule of venetoclax with AZD2811 dosing on Days 1, 4, 15 and 18 (see below) may be explored.

Group 3 Arm B will not exceed the registered venetoclax dose when combined with a starting dose of AZD2811 that is considered safe based on Group 3 Arm A observations. Subsequent cohorts will explore how to escalate AZD2811 in a more intensified schedule towards a recommended Phase 2 dose.

Part B - Dose Expansion

In Part B approximately 18 AML participants (6 additional participants in each group [AZD2811 monotherapy, Group 1], [AZD2811 in the azacitidine combination setting, Group 2], and [AZD2811 and venetoclax combination, Group 3]) will follow the affiliated dose/schedule from Part A that was found to be the most tolerable and/or efficacious.

ELIGIBILITY:
Inclusion criteria

1. AML participants who have either: (a) relapsed or are refractory to standard therapies (the participant may have been treated with standard therapy prior to the diagnosis of AML e.g. for MDS), OR (b) diagnosis of AML (bone marrow blasts ≥ 20%), who are previously untreated for AML, and are not suitable for intensive induction therapy, as defined below (for AZD2811 monotherapy and HMA combination participants only i.e. inclusion criteria 1(b) may only be used to enrol a participant into Groups 1 and 2; previously untreated AML participants may not enrol into Group 3 unless they fulfil inclusion criteria 1(a) above).

   Participants are unsuitable for intensive induction therapy if they are:
   * 75 years or

     * 75 years of age with clinically significant cardiac or pulmonary dysfunction unrelated to leukaemia, as reflected by at least 1 of the following criteria: Left ventricular ejection fraction (LVEF) ≤50% Diffusing capacity of the lungs for carbon monoxide (DLCO) ≤65% of expected Forced expiratory volume 1(FEV1) ≤65% of expected Chronic stable angina any significant co-morbidities which in the opinion of the treating physician makes the participant unsuitable for intensive induction therapy. This must be documented by the study monitor.
2. AML participants who are unlikely to demonstrate rapid progression such that they would be unable to complete the first cycle of therapy.
3. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling and analyses.
4. Aged at least 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
6. Prior treatment with hydroxyurea (up to 24 hours before study treatment) is allowed
7. Adequate organ system function as outlined below:

   Prothrombin time (PT)/partial thromboplastin time (PTT) ≤1.5 x upper limit of normal (ULN) Total bilirubin ≤1.5 x ULN. Participants with documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) who have serum bilirubin ≤3 x the ULN may be enrolled, unless there is evidence of hemolytic anemia Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ˂2.5 x ULN if no liver involvement or ≤5 times the ULN with liver involvement Creatinine ≤1.5 x ULN, OR calculated or measured creatinine clearance ≥50 mL/min as calculated by the Cockcroft-Gault method, OR 24-hour measured urine creatinine clearance ≥50 mL/min.

   Participants enrolled in the venetoclax combination part with a creatinine clearance (CLcr) <80 mL/min (and ≥ 45 mL/min) as calculated by Cockcroft-Gault should be able to have more intensive prophylaxis and monitoring (according to institutional standard) to reduce the risk of tumour lysis syndrome (TLS) when initiating treatment with venetoclax.
8. Females should be using adequate contraception, should not be breast feeding and must have a negative serum pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: a) Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments, b) have documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

9 Sexually active male participants should be willing to use barrier contraception i.e., condoms. Female partners of male participants should also use a highly effective form of contraception if they are of childbearing potential, unless the male participant is abstaining from sexual intercourse.

Exclusion criteria

1. Treatment with any of the following:

   Any investigational agents, experimental antibody or antibody drug conjugates, or study drugs from a previous clinical study within 3-4 weeks of said prior investigational agent(s) with regard to the first dose of study treatment on this clinical study protocol.

   Any other chemotherapy (except hydroxyurea), immunotherapy or anticancer agents within 2 weeks of the first dose of study treatment

   Any haematopoietic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) within 7 days of the first dose of AZD2811 monotherapy or with combination agent(s) or pegylated G-CSF (pegfilgrastim) or darbepoetin within 14 days of the first dose of study treatment

   Prescription or non-prescription drugs or other products known to be strong inhibitors/inducers of CYP3A that cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug. Washout periods should be a minimum of 5 half-lives depending on the medication.

   Participants who have undergone allogeneic stem cell transplant within 12 months are excluded. If allogeneic transplant was >12 months ago, then they are not excluded as long as they are off all immunosuppression and have no signs or symptoms of active graft versus host disease.

   Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
2. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment .
3. Presence of, or history of leptomeningeal disease.
4. As judged by the Investigator, any evidence of: severe or uncontrolled systemic diseases (e.g., severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]) or other malignancy (like advanced malignant hepatic tumours); current unstable or uncompensated respiratory or cardiac conditions; or uncontrolled hypertension; history of, or active, bleeding diatheses (e.g., haemophilia or von Willebrand disease); participants with inflammatory bowel disease (e.g., Crohn or colitis ulcerosa); uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment); or IV anti-infective treatment within 2 weeks before first dose of study treatment unless either clear evidence would indicate that despite the clinical symptoms no infection took place, or just a single dose of IV antibiotics was administered followed by oral treatment thereafter.
5. Any of the following cardiac criteria: a) Congestive heart failure (CHF) per New York Heart Association (NYHA) classification > Class II, b) Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, c) Unstable angina or new-onset angina, d) QTcF interval >450 ms (for male participants) or >470 ms (for female participants) on screening electrocardiogram (ECG).
6. Active non-infectious skin disease (including rash, dermatitis, or psoriasis, but excluding stable plaque psoriasis from the definition of active disease). Participants with a rash that is biopsy-proven leukaemia or with pressure ulcers are not excluded. Participants with petechiae from thrombocytopenia or participants with drug related rashes that are improving are not excluded..
7. Participants with a known hypersensitivity to azacitidine or mannitol (HMA combination participants only).
8. History of hypersensitivity to active or inactive excipients (e.g., PEG) of any drug in the study or drugs with a similar chemical structure or class to those investigated in the study.
9. Known history of infection with human immunodeficiency virus (HIV)
10. Serologic status reflecting active hepatitis B or C infection:

    1. Participants who are anti-HBc positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result before enrolment. Those who are hepatitis B surface antigen positive or hepatitis B PCR positive will be excluded.
    2. Participants who are hepatitis C antibody positive will need to have a negative PCR result before enrolment. Those who are hepatitis C PCR positive will be excluded.

Additional exclusion criteria - venetoclax combination

1. Adults with previously untreated diagnosis of AML (bone marrow blasts ≥ 20%), unless they fulfil inclusion criterion 1(a) above.
2. White blood cell (WBC) count > 25,000 cells/mm^3 (25 x 10^9/L); use of leukapheresis or hydroxyurea before venetoclax initiation is allowed to achieve this entry criterion (leukapheresis or hydroxyurea must be stopped at least 48 hours before the initiation of venetoclax).
3. AML with known active central nervous system involvement.
4. Chronic respiratory disease that requires continuous oxygen use.
5. Previous venetoclax exposure that ended due to venetoclax toxicity.
6. Use of moderate CYP3A inhibitor/inducers and P-gP inhibitors, with the exception of fluconazole and isavuconazole, that cannot be discontinued prior to Day 1 of dosing. Washout periods should be a minimum of 5 half-lives depending on the medication unless agreed upon with the Sponsor.
7. Participant consumed grapefruit, grapefruit products, Seville oranges (including marmalades containing Seville oranges) or star fruit within 3 days before the initiation of venetoclax.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) | Day 1 to Day 28 of first cycle
  A DLT was defined as any adverse event (AE) not related to the underlying leukaemia requiring treatment interruption for > 21 days, any Grade 5 AE, Grade 4 neutropenia or thrombocytopenia lasting >= 42 days from start of cycle in absence of evidence of active leukaemia, any >= Grade 3 non-haematological AE (except Grade 3 nausea, vomiting, mucositis, stomatitis or diarrhoea that was controlled within 4 days and Grade 3 elevations in alanine aminotransferase/ aspartate aminotransferase that return to meet initial eligibility criteria within 7 days of study drug interruption), or any other clinically significant and/or unacceptable AE that does not respond to supportive care, results in a disruption of dosing schedule for > 7 days, or was judged as a DLT by Investigator in collaboration with the Medical Monitor. An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Day 1 through early termination of the study (approximately 42 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. There will be no updated results for this outcome measures at the time of end of study.
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Grade 4 TEAEs | Day 1 through early termination of the study (approximately 42 months)
  Participants with abnormal clinical laboratory parameters reported as Grade 4 TEAEs are reported. Laboratory analysis included hematology, clinical chemistry, and urinalysis.
  hematology, coagulation, chemistry, and urinalysis parameters over time are reported.

SECONDARY OUTCOMES:
Number of Participants With Total Complete Remission (CR) | Day 1 through early termination of the study (approximately 42 months)
  Total complete remission included CR and CR with incomplete recovery (CRi). The CR is defined as bone marrow blasts <5%, absence of blasts with Auer rods, absence of extramedullary disease, absolute neutrophil count >1.0 × 10/L, platelet count >100 × 10/L, and independence of red cell transfusions. The CRi includes all CR criteria except for residual neutropenia (<1.0 × 10/L) or thrombocytopenia (<100 × 10/L).
Number of Participants With Overall Response Rate (ORR) | Day 1 through early termination of the study (approximately 42 months)
  The ORR included CR, CRi, and partial remission (PR). The CR is defined as bone marrow blasts <5%, absence of blasts with Auer rods, absence of extramedullary disease, absolute neutrophil count >1.0 × 10/L, platelet count >100 × 10/L, and independence of red cell transfusions. The CRi includes all CR criteria except for residual neutropenia (<1.0 × 10/L) or thrombocytopenia (<100 × 10/L). The PR is defined as all hematologic criteria of CR (absolute neutrophil count >1.0 × 10/L, platelet count >100 × 10/L, and independence of red cell transfusions), decrease of bone marrow blast percentage to 5% to 25%, and decrease of pre-treatment bone marrow blast percentage by at least 50%.
Number of Participants With Partial Remission (PR) | Day 1 through early termination of the study (approximately 42 months)
  The PR is defined as all hematologic criteria of CR (absolute neutrophil count >1.0 × 10/L, platelet count >100 × 10/L, and independence of red cell transfusions), decrease of bone marrow blast percentage to 5% to 25%, and decrease of pre-treatment bone marrow blast percentage by at least 50%.
Number of Participants With >50% Change in Bone Marrow Blasts from Baseline in Participants With AML | Baseline (Day 1), Cycle 1 Day 22, Cycle 2 Day 22, Cycle 4 Day 22, and end of treatment (approximately 42 months)
  Participants with >50% change in myleloblasts from baseline are reported.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (11):
- United States (10):
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Detroit, Michigan
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Research Site, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6130C00003&attachmentIdentifier=e3ca00bb-7b92-41e9-b56c-c7079c2d691d&fileName=d6130c00003_CSRSynopsis.pdf&versionIdentifier=